CLINICAL TRIAL: NCT05084794
Title: Does Fixation of Medium-sized Posterior Malleolus Fractures Provide Better Outcome?
Brief Title: The Results of Middle-sized Posterior Malleolus Fractures: Fixed Versus Non-fixed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Bedri Karaismailoglu, Assistant Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-22/01.09.2015
Record Dates: First submitted 2021-10-08; First posted 2021-10-20 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Ankle Fractures; Posterior Malleolus Fractures
Keywords: ankle; fracture; posterior; malleolus; fixation
MeSH Terms: conditions — Ankle Fractures; Fractures, Bone | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-fixated (No Intervention): Posterior malleolus fractures won't be fixated.
- Fixated (Experimental): Posterior malleolus fractures will be fixated with either plate or screws.
  Interventions: Procedure: Internal fixation

INTERVENTIONS:
Procedure: Internal fixation — Fixation of posterior malleolus with either plate or screws.
  Arms: Fixated

SUMMARY:
This study aims prospective randomized comparison of mid-term clinical outcomes of middle-sized posterior malleolus fractures with and without internal fixation.

DETAILED DESCRIPTION:
Although it has traditionally been accepted that posterior malleolar fractures involving less than 25 percent of the tibial plafond do not require operative fixation, this belief is now questioned. A number of studies have shown that the posterior malleolus contributes significantly to ankle stability. Many studies have also demonstrated that postoperative outcomes are better in patients who underwent posterior malleolar reduction and fixation.

The aim of this prospective study is to show how internal fixation of the posterior malleolus, including middle-sized posterior malleolar fractures (10-25%), affects clinical outcomes and to discuss the factors that may lead to arthritis of the ankle joint. The groups will be randomized. The clinical and functional results of 40 patients who will be operated between 2015-2019 due to ankle fracture will be evaluated at short to mid-term (2-5 years). According to our hypothesis, internally fixed posterior malleolar fractures give better clinical and functional scores.

ELIGIBILITY:
Inclusion Criteria:

Patients who were operated for ankle fractures, including posterior malleolar fracture between 10-25% of the joint surface. Two to five years of follow-up with functional and radiological outcome.

Exclusion Criteria:

Posterior malleolar fractures accompanied by severe soft tissue damage after high-energy injury will not be included in the study. Written consent will be obtained from all participants, patients who do not give consent or refuse to participate will not be included in the study. Patients who left the study voluntarily will not be included in the statistics. Patients with additional joint disorders, previous surgery or previous history of ankle complaint will not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Short Musculoskeletal Function Assessment (SMFA) Questionnaire | 2 year
  Functional outcome score between 0 and 100. Higher score indicates a worse function.
Kellgren-Lawrence grading system for osteoarthritis | 2 year
  Grade of ankle osteroarthritis. Score between 0 to 4. Higher score indicates worse joint cartilage.
American Orhopaedic Foot and Ankle Score (AOFAS) Score | 5 year
  Functional outcome score between 0 and 100. Higher score indicates better function.

IPD SHARING:
Plan to Share IPD: No